CLINICAL TRIAL: NCT06583538
Title: An Online Rehabilitation Programme to Support Physical Activity Adherence and Functional Capacity in People with Spinal Cord Injury Following Discharge Into the Community: a Feasibility Study
Brief Title: An Online Rehabilitation Programme for People with SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 331702
Record Dates: First submitted 2023-12-15; First posted 2024-09-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injuries; Physical Inactivity; Spinal Cord Injury, Acute
MeSH Terms: conditions — Spinal Cord Injuries; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online Exercise (Experimental): Online personalised rehabilitation consisting of strengthening, aerobic and stretching. 40mins per session, twice per week, for 12 weeks
  Interventions: Other: Giraffe Healthcare

INTERVENTIONS:
Other: Giraffe Healthcare — An online personalised rehabilitation platform consisting of exercise videos with written and audio instruction, an exercise diary, advice and in-built messaging system between therapist and participant.
  The exercise prescription consists of strengthening, aerobic and stretching. 40mins per session, twice per week, for 12 weeks

SUMMARY:
The goal of this feasibility study is to explore the feasibility and effectiveness of a 12-week online rehabilitation programme in people with Spinal Cord Injury during the transition from hospital to home.

The main question[s] it aims to answer are:

* What is the feasibility of an online rehabilitation programme to support physical activity adherence in people with spinal cord injury following discharge into the community?
* How effective is an online rehabilitation programme to enhance functional capacity, physical activity and quality of life in people with spinal cord injury following discharge into the community?

Participants will be given a personalised online rehabilitation programme to complete two times a week. It will consist of a warm up two exercise components (cardiorespiratory fitness and muscle strength) and a cool down.

DETAILED DESCRIPTION:
Bridging the gap between the inpatient setting to the home environment is essential to promote Physical Activity (PA) adherence, improve functional independence and enhance quality of life by implementing lifelong exercise habits. To our knowledge, no study has investigated the feasibility of an online rehabilitation programme among sub-acute Spinal Cord Injury (SCI) patients during this important discharge period from hospital to home. Therefore, this study will explore the feasibility and effectiveness of a 12-week online rehabilitation programme in people with SCI during the transition from hospital to home.

All subacute inpatients who are undergoing their first episode of inpatient rehabilitation post SCI at the Queen Elizabeth National Spinal Injuries Unit (QENSIU) who fulfil the inclusion criteria will be invited to take part in the current study. A rehabilitation programme will be prescribed individually for each participant. Each programme will align with the current PA guidelines for adults with SCI and will be tailored to the participants ability. Participants will be advised to complete the programme twice per week. It will consist of 20 mins cardiorespiratory followed by a strengthening session. Therefore, the participants will engage in the programme for roughly 40 minutes twice per week. The participants will be instructed to log all completed sessions in an online diary so adherence and duration of PA can be monitored.

Assessment will consist of 4 phases, two in person assessments at baseline and 6 weeks post discharge and two remote (online) assessments at 2 and 12 weeks post discharge. Each assessment will consist of quantitative outcome measures. Additionally, a subset of the study sample will take part in a qualitative structured video interview at the end of their intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at the Queen Elizabeth National Spinal Injuries Unit
* Incomplete or complete spinal cord injury of less than one year in duration
* Medically stable to engage in physical rehabilitation and physical activity
* Able to engage in manual wheelchair propulsion and / or weight baring activities
* Discharge date anticipated within the next 4 weeks
* Access and capability to use the internet

Exclusion Criteria:

* Under 18 years old
* Chronic spinal cord injury patients more than one year since injury
* Discharge planned to another hospital or care facility
* Co-morbidities which would preclude taking part in a physical activity programme: medically diagnosed ischemic heart disease; unstable angina, dysrhythmia or unstable autonomic dysreflexia; recent osteoporotic fracture, tracheostomy, current pressure injury, current substance dependence, psychosis, severe chronic upper extremity pain, surgery pending within 6 months, recurrent infection or illness requiring hospitalization (Bombardier et al., 2021).
* Those who do not wish to take part in a physical activity research study
* Unable to understand written and spoken English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Adherence | 12 weeks
  Adherence will be monitored remotely by the number of online diary entries per participant.á Adherence will then be calculated based on percentage of completed sessions per week over the 12 weeks.Following the guidelines, the optimum number of completed sessions per participant is 2 x 20 mins cardiorespiratory and 2 strengthening per week. >75% = excellent , 50-75% = good, <50% = satisfactory, <25% = low.
Acceptability | Week 6 to week 12
  Acceptability will be captured by the structured online video interview. Thematic analysis will be used to assess the qualitative data.
Participant recruitment and retention | 12 weeks
  Measured by assessing participant eligibility (number of those approached and those who meet the inclusion criteria), recruitment rate per month and retention of recruited participants.

SECONDARY OUTCOMES:
Self-report Physical Activity Scale for individuals with Physical Disabilities (PASIPD) | Baseline, Week 2, Week 6 and week 12
  Captures information about leisure, household and work-related activity over the preceding 7 days.The PASIPD calculates scores by multiplying the time spent on each activity by a metabolic equivalent value (MET) and then adding the results together with a maximum score of 199.5. Individuals respond to 2 ordinally ranked responses. Frequency responses range from 1 (never) to 4 (often) while duration responses range from 1 (less than 1) hour to 4 (greater than 4 hours).
6-minute wheelchair test (6minWCT) OR 6-minute walk test (6MinWT) | Baseline and week 6
  Assesses functional capacity and endurance
Muscle Strength in kg | Baseline and week 6
  Via manual muscle dynamometer
Borg Rate of Perceived Exertion (RPE) Scale | Baseline and week 6
  Collected after 6 minute test. 6-20 point self-reported scale based on rate of perceived exertion with 6 being minimum and 20 being maximum.
Walking Index for Spinal Cord Injury (WISCI II) | Baseline and week 6
  Assesses improvement in walking ability. Measures type and level of assistance required for walking 10m. Minimum = 0, Maximum = 20.
Spinal Cord Independence Measure Self Report (SCIM III SR) | Baseline, Week 2, Week 6 and week 12
  Performance in activities of daily living and mobility questionnaire.The SCIM-SR assesses the degree of independence an individual with SCI has in 3 categories; self-care, respiration and sphincter management and mobility. A higher score indicates greater functional independence. Maximum = 100.
World Health Organisation Quality of Life-Bref Scale (WHOQoL-Bref) | Baseline, Week 2, Week 6 and week 12
  Quality of life questionnaire measures 4 domains: physical, psychological, social and environmental health. Higher score indicates greater quality of life. Maximum = 400.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Coulter, PhD, Study Chair — Glasgow Caledonian University
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, Scotland, United Kingdom